CLINICAL TRIAL: NCT04201327
Title: Unified Approach to Address PrEP Care Cascade
Brief Title: Project Jumpstart for Improving PrEP Care of Continuum Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lisa Eaton, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H17-335; R34MH115798 (NIH)
Record Dates: First submitted 2019-11-25; First posted 2019-12-17 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: 4 arm randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator and the assessment staff are blind to the assignment of participants throughout the data collection phase of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PrEP information only arm (Active Comparator): Information to for accessing HIV prevention tools will be provided to participants.
  Interventions: Behavioral: Project Jumpstart
- PrEP counseling arm (Experimental): Stigma focused counseling (one-session) aimed at addressing barriers to health care access will be provided.
  Interventions: Behavioral: Project Jumpstart
- PrEP counseling plus text messaging arm (Experimental): Stigma focused counseling (one-session) and interactive text messaging aimed at addressing barriers to health care access will be provided.
  Interventions: Behavioral: Project Jumpstart
- PrEP counseling plus text messaging and on demand counseling (Experimental): Ongoing stigma focused counseling and interactive text messaging aimed at addressing barriers to health care access will be provided.
  Interventions: Behavioral: Project Jumpstart

INTERVENTIONS:
Behavioral: Project Jumpstart — PrEP focused intervention to improve PrEP related health outcomes

SUMMARY:
Stigma related to PrEP interest and uptake, and medication cognitions related to PrEP adherence and persistence remain strong barriers to improving PrEP use. To address these areas, the investigators are proposing to develop an intervention grounded in two novel cognitive/behavioral theories: the HIV Stigma Framework and the Medication Necessity-Concerns Framework. Advances in biomedical HIV prevention, such as the availability of PrEP, will only impact the HIV epidemic if concurrent efforts are made to address the social and behavioral challenges that are associated with achieving sufficient coverage of PrEP among individuals at elevated risk for HIV.

DETAILED DESCRIPTION:
Biomedical HIV prevention tools are very promising, but are not sufficiently reaching those in greatest need. BMSM have experienced elevated rates of HIV incidence and prevalence since the beginning of the US epidemic, and the CDC estimates that half of BMSM will be diagnosed with HIV in their lifetime. Although Pre-Exposure Prophylaxis (PrEP) is highly effective for preventing HIV, there is urgent need to improve efforts to deliver PrEP, in particular, for BMSM at-risk for HIV. Current strategies to increase PrEP interest, uptake, and adherence are not adequate and there are formidable barriers (e.g., stigma surrounding PrEP use, and adherence and retention concerns) to sufficient coverage of PrEP that must be addressed. Without considerable and targeted change to our current approach to PrEP delivery, public health initiatives will fail to adequately provide PrEP to those in greatest need. In our PrEP focused preliminary studies with BMSM, the investigators have identified two primary areas in need of critical focus and intervention - (1) stigma related to PrEP use, and (2) medication cognitions such as the perceived costs and benefits of taking PrEP, both of which can impede PrEP interest, uptake, and adherence. To address these areas the investigators have developed an intervention grounded in two novel cognitive/behavioral theories: the HIV Stigma Framework and the Medication Necessity-Concerns Framework. Our study includes: Conducting a pilot test that compares our (a) PrEP information only control (n=25), (b) PrEP counseling (n=50), (c) PrEP counseling with text messages (n=50), and (d) PrEP enhancement counseling with text messaging and on-demand counseling (n=50). Advances in biomedical HIV prevention, such as the availability of PrEP, will only impact the HIV epidemic if concurrent efforts are made to address the social and behavioral challenges that are associated with achieving sufficient coverage of PrEP among individuals at elevated risk for HIV. Low-resource burden, easily implemented, and effective social/behavioral interventions are urgently needed if the full benefits of PrEP are to be realized. If effective and disseminated, this intervention would meet current prevention needs and its potential impact on HIV infections averted could be substantial.

ELIGIBILITY:
Inclusion Criteria:

* Prior sex with a man, identify as Black, and HIV negative status.

Exclusion Criteria:

* Living with HIV

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
PrEP Linkage | 6 months
  Number of participants who attend PrEP care appointment. Documentation will be provided from clinic.
PrEP Uptake | 6 months
  Number of participants who receive PrEP prescription from provider. Documentation will be provided from clinic.
PrEP Adherence | 6 months
  Number of participants who adhere to PrEP medications. Documentation will be provided through self report and urine tests (UrSure).

CONTACTS AND LOCATIONS:
Locations (1):
- SHARE Project, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eaton LA, Layland EK, Driver R, Kalichman SC, Kalichman MO, Watson RJ, Kalinowski J, Chandler CJ, Earnshaw VA. Novel Latent Profile Analysis of a Test of Concept, Stigma Intervention to Increase PrEP Uptake Among Black Sexual Minority Men. J Acquir Immune Defic Syndr. 2023 Sep 1;94(1):1-9. doi: 10.1097/QAI.0000000000003223. PMID 37195906